CLINICAL TRIAL: NCT02840045
Title: Development of a New Neuroimaging Method Aimed to Differentiate Mnesic Abilities of Alzheimer and Depressed Patients
Acronym: RIHANNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: API/2014/51
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer Disease; Depression
Keywords: electroencephalography (EEG)
MeSH Terms: conditions — Alzheimer Disease; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alzheimer patients (Experimental): Cerebral measurements from high-density electroencephalography are recorded in Alzheimer patients. The same protocol is applied in the 3 arms
  Interventions: Device: high-density electroencephalography
- patients with a depressive disorder (Experimental): Cerebral measurements from high-density electroencephalography are recorded in patients with a depressive disorder. The same protocol is applied in the 3 arms
  Interventions: Device: high-density electroencephalography
- Healthy controls (Active Comparator): Cerebral measurements from high-density electroencephalography are recorded in healthy controls
  Interventions: Device: high-density electroencephalography

INTERVENTIONS:
Device: high-density electroencephalography — Musical stimulation during electroencephalography recording

SUMMARY:
The purpose of this study is to use a new method to differentiate mnesic abilities of early alzheimer patients and patients with a depressive disorder.

This method is based on the recording of cerebral activity while patients listen to familiar, unfamiliar and newly-learned music.

ELIGIBILITY:
Inclusion Criteria:

* Being right-handed
* recorded consent
* For Alzheimer patients: Mini Mental Status Examination (MMSE) score >= 18
* For patients with a depressive disorder : Major Depressive Disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM IV) and Montgomery-Asberg depression rating scale (MADRS) score >= 25
* For healthy controls : no cognitive deficit, MADRS score < 25, no depressive disorder according to DSM IV

Exclusion Criteria:

* Auditory deficit
* contraindication to a high-density electroencephalography exam
* refusal to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02-20 (Actual); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-08-20 (Estimated)

PRIMARY OUTCOMES:
Amplitude of event-related potentials | day 1 for familiar and unfamiliar songs and day 14 for newly learned songs
  Measurements of the amplitude of event-related potentials with electroencephalography at day one for familiar and unfamiliar songs and after 2 weeks for newly learned songs

SECONDARY OUTCOMES:
Spectral power | day 1 for familiar and unfamiliar songs and day 14 for newly learned songs
  Measurements of the spectral power with electroencephalography at day one for familiar and unfamiliar songs and after 2 weeks for newly learned songs

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vandel, MD, PhD, Principal Investigator — Service de psychiatrie
Locations (1):
- CHRU Besançon, Besançon, Franche-Comte, France

REFERENCES:
- [Background] Gabriel D, Wong TC, Nicolier M, Giustiniani J, Mignot C, Noiret N, Monnin J, Magnin E, Pazart L, Moulin T, Haffen E, Vandel P. Don't forget the lyrics! Spatiotemporal dynamics of neural mechanisms spontaneously evoked by gaps of silence in familiar and newly learned songs. Neurobiol Learn Mem. 2016 Jul;132:18-28. doi: 10.1016/j.nlm.2016.04.011. Epub 2016 Apr 27. PMID 27131744